CLINICAL TRIAL: NCT00466336
Title: Prediction of Hepatic Fibrosis in Patients With Chronic Hepatitis C by Biochemical and Duplex Doppler Indices
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 200612012R
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-03

CONDITIONS: Chronic Hepatitis C; Hepatic Fibrosis; Cirrhosis
Keywords: Chronic hepatitis C; Non-invasive diagnosis; Duplex Doppler ultrasonography; Biochemical indices; Hepatic fibrosis; Cirrhosis
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of our prospective study was to evaluate the value of Doppler parameters and compare the diagnostic accuracy of Doppler parameters with various biochemical indices in predicting significant hepatic fibrosis (≥ F2) and cirrhosis (F4) in chronic hepatitis C (CHC) patients.

DETAILED DESCRIPTION:
Chronic hepatitis C virus (HCV) infection is a global health problem, affecting about 3% of the world's population. Compared to patients with mild hepatic fibrosis, those with significant fibrosis are at risk of developing cirrhosis over a 10- to 20-year period. This fact suggests the need of early antiviral therapy in chronic hepatitis C (CHC) patients to prevent the development of cirrhosis and associated complications. For patients having cirrhosis, surveillance endoscopy and ultrasound for gastroesophageal varices and hepatocellular carcinoma are needed to minimize morbidity and mortality ). Furthermore, reduced treatment response and tolerability to antiviral therapy may be encountered in cirrhotic patients. An accurate assessment of hepatic fibrosis stage is therefore important for both diagnostic and therapeutic purposes.

Liver biopsy has been recognized as the gold standard for assessing the grade of necroinflammation and stage of fibrosis. However, it is costly, and harbors risk of complications, including 20% of patient discomfort, 0.1-3% of significant morbidity, and 0.02-0.24% of mortality. In addition, sampling error due to the non-uniform distribution of the parenchymal damage, as well as intra- and inter-observer variability is often encountered. A noninvasive tool to evaluate liver disease activity or fibrosis stage would be helpful, particularly in monitoring CHC patients over time.

Noninvasive methods to evaluate the hepatic histology in HCV-infected patients include symptoms and signs, routine laboratory tests, serum markers of fibrosis and inflammation, quantitative tests of liver function, and radiological imaging. Previous studies have assessed the usefulness of noninvasive tests in predicting hepatic fibrosis. However, none of them showed satisfactory results, either due to lack of accuracy, accessibility, reproducibility or being expensive.

Duplex Doppler ultrasonography (DDU), which is readily available and non-invasive, has been used for the assessment of splanchnic vascular hemodynamics in patients with chronic liver disease. Portal vein velocity (PVV) has been shown to be correlated with significant fibrosis or cirrhosis. Hepatic artery resistive index (HARI) and pulsatility index (HAPI) are associated with portal vein resistance and hepatic vein-portal vein pressure gradient (HPVG). Splenic artery resistive index (SARI) and pulsatility index (SAPI) are associated with portal vein resistance, cirrhosis and grade of esophageal varices (EV). Previous studies to evaluate the value of DDU in predicting liver histology are controversial, probably due to small patient number, diverse grading of liver histology, and large missing data.

Thus, the purpose of our prospective study was to evaluate the value of Doppler parameters and compare the diagnostic accuracy of Doppler parameters with various biochemical indices in predicting significant hepatic fibrosis (≥ F2) and cirrhosis (F4) in chronic hepatitis C (CHC) patients.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Positive anti-HCV and HCV RNA for more than 6 months
* Alanine aminotransferase level more than twice the upper limit of normal (ULN)

Exclusion Criteria:

* HBV and HCV co-infection
* HIV and HCV co-infection
* Heavy alcohol use (> 50 gram/day)
* Autoimmune liver diseases
* Metabolic liver diseases
* Presence of hepatocellular carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis C patients with abnormal ALT levels (> 2X ULN) with percutaneous liver biopsy
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2003-01; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, Study Director — Department of Internal Medicine, National Taiwan Universitys Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] National Institutes of Health Consensus Development Conference Panel statement: management of hepatitis C. Hepatology. 1997 Sep;26(3 Suppl 1):2S-10S. doi: 10.1002/hep.510260701. PMID 9305656
- [Background] Lauer GM, Walker BD. Hepatitis C virus infection. N Engl J Med. 2001 Jul 5;345(1):41-52. doi: 10.1056/NEJM200107053450107. No abstract available. PMID 11439948
- [Background] Yano M, Kumada H, Kage M, Ikeda K, Shimamatsu K, Inoue O, Hashimoto E, Lefkowitch JH, Ludwig J, Okuda K. The long-term pathological evolution of chronic hepatitis C. Hepatology. 1996 Jun;23(6):1334-40. doi: 10.1002/hep.510230607. PMID 8675148
- [Background] de Franchis R, Pascal JP, Ancona E, Burroughs AK, Henderson M, Fleig W, Groszmann R, Bosch J, Sauerbruch T, Soederlund C, et al. Definitions, methodology and therapeutic strategies in portal hypertension. A Consensus Development Workshop, Baveno, Lake Maggiore, Italy, April 5 and 6, 1990. J Hepatol. 1992 May;15(1-2):256-61. doi: 10.1016/0168-8278(92)90044-p. No abstract available. PMID 1506645
- [Background] Daniele B, Bencivenga A, Megna AS, Tinessa V. Alpha-fetoprotein and ultrasonography screening for hepatocellular carcinoma. Gastroenterology. 2004 Nov;127(5 Suppl 1):S108-12. doi: 10.1053/j.gastro.2004.09.023. PMID 15508073
- [Background] Heathcote EJ, Shiffman ML, Cooksley WG, Dusheiko GM, Lee SS, Balart L, Reindollar R, Reddy RK, Wright TL, Lin A, Hoffman J, De Pamphilis J. Peginterferon alfa-2a in patients with chronic hepatitis C and cirrhosis. N Engl J Med. 2000 Dec 7;343(23):1673-80. doi: 10.1056/NEJM200012073432302. PMID 11106716
- [Background] Piccinino F, Sagnelli E, Pasquale G, Giusti G. Complications following percutaneous liver biopsy. A multicentre retrospective study on 68,276 biopsies. J Hepatol. 1986;2(2):165-73. doi: 10.1016/s0168-8278(86)80075-7. PMID 3958472
- [Background] Nord HJ. Biopsy diagnosis of cirrhosis: blind percutaneous versus guided direct vision techniques--a review. Gastrointest Endosc. 1982 May;28(2):102-4. doi: 10.1016/s0016-5107(82)73015-9. No abstract available. PMID 6211383
- [Background] Garcia-Tsao G, Boyer JL. Outpatient liver biopsy: how safe is it? Ann Intern Med. 1993 Jan 15;118(2):150-3. doi: 10.7326/0003-4819-118-2-199301150-00013. No abstract available. PMID 8416312
- [Background] Cadranel JF, Rufat P, Degos F. Practices of liver biopsy in France: results of a prospective nationwide survey. For the Group of Epidemiology of the French Association for the Study of the Liver (AFEF). Hepatology. 2000 Sep;32(3):477-81. doi: 10.1053/jhep.2000.16602. PMID 10960438
- [Background] McGill DB, Rakela J, Zinsmeister AR, Ott BJ. A 21-year experience with major hemorrhage after percutaneous liver biopsy. Gastroenterology. 1990 Nov;99(5):1396-400. doi: 10.1016/0016-5085(90)91167-5. PMID 2101588
- [Background] Maharaj B, Maharaj RJ, Leary WP, Cooppan RM, Naran AD, Pirie D, Pudifin DJ. Sampling variability and its influence on the diagnostic yield of percutaneous needle biopsy of the liver. Lancet. 1986 Mar 8;1(8480):523-5. doi: 10.1016/s0140-6736(86)90883-4. PMID 2869260
- [Background] Bedossa P, Dargere D, Paradis V. Sampling variability of liver fibrosis in chronic hepatitis C. Hepatology. 2003 Dec;38(6):1449-57. doi: 10.1016/j.hep.2003.09.022. PMID 14647056
- [Background] Colloredo G, Guido M, Sonzogni A, Leandro G. Impact of liver biopsy size on histological evaluation of chronic viral hepatitis: the smaller the sample, the milder the disease. J Hepatol. 2003 Aug;39(2):239-44. doi: 10.1016/s0168-8278(03)00191-0. PMID 12873821
- [Background] Fontana RJ, Lok AS. Noninvasive monitoring of patients with chronic hepatitis C. Hepatology. 2002 Nov;36(5 Suppl 1):S57-64. doi: 10.1053/jhep.2002.36800. PMID 12407577
- [Background] Williams AL, Hoofnagle JH. Ratio of serum aspartate to alanine aminotransferase in chronic hepatitis. Relationship to cirrhosis. Gastroenterology. 1988 Sep;95(3):734-9. doi: 10.1016/s0016-5085(88)80022-2. PMID 3135226
- [Background] Sheth SG, Flamm SL, Gordon FD, Chopra S. AST/ALT ratio predicts cirrhosis in patients with chronic hepatitis C virus infection. Am J Gastroenterol. 1998 Jan;93(1):44-8. doi: 10.1111/j.1572-0241.1998.044_c.x. PMID 9448172
- [Background] Park GJ, Lin BP, Ngu MC, Jones DB, Katelaris PH. Aspartate aminotransferase: alanine aminotransferase ratio in chronic hepatitis C infection: is it a useful predictor of cirrhosis? J Gastroenterol Hepatol. 2000 Apr;15(4):386-90. doi: 10.1046/j.1440-1746.2000.02172.x. PMID 10824882
- [Background] Giannini E, Risso D, Botta F, Chiarbonello B, Fasoli A, Malfatti F, Romagnoli P, Testa E, Ceppa P, Testa R. Validity and clinical utility of the aspartate aminotransferase-alanine aminotransferase ratio in assessing disease severity and prognosis in patients with hepatitis C virus-related chronic liver disease. Arch Intern Med. 2003 Jan 27;163(2):218-24. doi: 10.1001/archinte.163.2.218. PMID 12546613
- [Background] Imbert-Bismut F, Ratziu V, Pieroni L, Charlotte F, Benhamou Y, Poynard T; MULTIVIRC Group. Biochemical markers of liver fibrosis in patients with hepatitis C virus infection: a prospective study. Lancet. 2001 Apr 7;357(9262):1069-75. doi: 10.1016/S0140-6736(00)04258-6. PMID 11297957
- [Background] Myers RP, Ratziu V, Imbert-Bismut F, Charlotte F, Poynard T; MULTIVIRC Group. Groupe d'Etude Multidisciplinaire sur les Pathologies Liees au Virus C. Biochemical markers of liver fibrosis: a comparison with historical features in patients with chronic hepatitis C. Am J Gastroenterol. 2002 Sep;97(9):2419-25. doi: 10.1111/j.1572-0241.2002.05997.x. PMID 12358267
- [Background] Poynard T, Bedossa P. Age and platelet count: a simple index for predicting the presence of histological lesions in patients with antibodies to hepatitis C virus. METAVIR and CLINIVIR Cooperative Study Groups. J Viral Hepat. 1997 May;4(3):199-208. doi: 10.1046/j.1365-2893.1997.00141.x. PMID 9181529
- [Background] Wai CT, Greenson JK, Fontana RJ, Kalbfleisch JD, Marrero JA, Conjeevaram HS, Lok AS. A simple noninvasive index can predict both significant fibrosis and cirrhosis in patients with chronic hepatitis C. Hepatology. 2003 Aug;38(2):518-26. doi: 10.1053/jhep.2003.50346. PMID 12883497
- [Background] Forns X, Ampurdanes S, Llovet JM, Aponte J, Quinto L, Martinez-Bauer E, Bruguera M, Sanchez-Tapias JM, Rodes J. Identification of chronic hepatitis C patients without hepatic fibrosis by a simple predictive model. Hepatology. 2002 Oct;36(4 Pt 1):986-92. doi: 10.1053/jhep.2002.36128. PMID 12297848
- [Background] Castera L, Vergniol J, Foucher J, Le Bail B, Chanteloup E, Haaser M, Darriet M, Couzigou P, De Ledinghen V. Prospective comparison of transient elastography, Fibrotest, APRI, and liver biopsy for the assessment of fibrosis in chronic hepatitis C. Gastroenterology. 2005 Feb;128(2):343-50. doi: 10.1053/j.gastro.2004.11.018. PMID 15685546
- [Background] Lackner C, Struber G, Liegl B, Leibl S, Ofner P, Bankuti C, Bauer B, Stauber RE. Comparison and validation of simple noninvasive tests for prediction of fibrosis in chronic hepatitis C. Hepatology. 2005 Jun;41(6):1376-82. doi: 10.1002/hep.20717. PMID 15915455
- [Background] Rosenberg WM, Voelker M, Thiel R, Becka M, Burt A, Schuppan D, Hubscher S, Roskams T, Pinzani M, Arthur MJ; European Liver Fibrosis Group. Serum markers detect the presence of liver fibrosis: a cohort study. Gastroenterology. 2004 Dec;127(6):1704-13. doi: 10.1053/j.gastro.2004.08.052. PMID 15578508
- [Background] Gaiani S, Gramantieri L, Venturoli N, Piscaglia F, Siringo S, D'Errico A, Zironi G, Grigioni W, Bolondi L. What is the criterion for differentiating chronic hepatitis from compensated cirrhosis? A prospective study comparing ultrasonography and percutaneous liver biopsy. J Hepatol. 1997 Dec;27(6):979-85. doi: 10.1016/s0168-8278(97)80140-7. PMID 9453422
- [Background] Koda M, Murawaki Y, Kawasaki H, Ikawa S. Portal blood velocity and portal blood flow in patients with chronic viral hepatitis: relation to histological liver fibrosis. Hepatogastroenterology. 1996 Jan-Feb;43(7):199-202. PMID 8682462
- [Background] Sacerdoti D, Merkel C, Bolognesi M, Amodio P, Angeli P, Gatta A. Hepatic arterial resistance in cirrhosis with and without portal vein thrombosis: relationships with portal hemodynamics. Gastroenterology. 1995 Apr;108(4):1152-8. doi: 10.1016/0016-5085(95)90214-7. PMID 7698583
- [Background] Schneider AW, Kalk JF, Klein CP. Hepatic arterial pulsatility index in cirrhosis: correlation with portal pressure. J Hepatol. 1999 May;30(5):876-81. doi: 10.1016/s0168-8278(99)80142-1. PMID 10365815
- [Background] Bolognesi M, Sacerdoti D, Merkel C, Gerunda G, Maffei-Faccioli A, Angeli P, Jemmolo RM, Bombonato G, Gatta A. Splenic Doppler impedance indices: influence of different portal hemodynamic conditions. Hepatology. 1996 May;23(5):1035-40. doi: 10.1002/hep.510230515. PMID 8621130
- [Background] Bolognesi M, Sacerdoti D, Merkel C, Bombonato G, Gatta A. Noninvasive grading of the severity of portal hypertension in cirrhotic patients by echo-color-Doppler. Ultrasound Med Biol. 2001 Jul;27(7):901-7. doi: 10.1016/s0301-5629(01)00370-2. PMID 11476922
- [Background] Piscaglia F, Gaiani S, Calderoni D, Donati G, Celli N, Gramantieri L, Crespi C, Bolondi L. Influence of liver fibrosis on hepatic artery Doppler resistance index in chronic hepatitis of viral origin. Scand J Gastroenterol. 2001 Jun;36(6):647-52. doi: 10.1080/003655201750163178. PMID 11424325
- [Background] Lim AK, Patel N, Eckersley RJ, Kuo YT, Goldin RD, Thomas HC, Cosgrove DO, Taylor-Robinson SD, Blomley MJ. Can Doppler sonography grade the severity of hepatitis C-related liver disease? AJR Am J Roentgenol. 2005 Jun;184(6):1848-53. doi: 10.2214/ajr.184.6.01841848. PMID 15908541
- [Background] Aube C, Winkfield B, Oberti F, Vuillemin E, Rousselet MC, Caron C, Cales P. New Doppler ultrasound signs improve the non-invasive diagnosis of cirrhosis or severe liver fibrosis. Eur J Gastroenterol Hepatol. 2004 Aug;16(8):743-51. doi: 10.1097/01.meg.0000108357.41221.e5. PMID 15256975